CLINICAL TRIAL: NCT04552197
Title: A Phase 1, Open-Label, Multi-Dose Study to Assess the Systemic and Local Tissue Pharmacokinetics and Pharmacodynamics of JNJ-64251330 in Healthy Participants
Brief Title: A Study of JNJ-64251330 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR108808; 2020-000167-24 (EudraCT Number); 64251330EDI1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-08-28; First posted 2020-09-17 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1: Treatment A (JNJ-64251330) (Experimental): Participants will receive JNJ-64251330 (dose 1), once daily for 5 days under fasting conditions.
  Interventions: Drug: JNJ-64251330
- Part 1: Treatment B (JNJ-64251330) (Experimental): Participants will receive JNJ-64251330 (dose 1), twice daily for 5 days under fasting conditions.
  Interventions: Drug: JNJ-64251330
- Part 1: Treatment C (JNJ-64251330) (Experimental): Participants will receive JNJ-64251330 (dose 2), twice daily for 5 days under fasting conditions.
  Interventions: Drug: JNJ-64251330
- Part 1: Treatment D (JNJ-64251330) (Active Comparator): Participants will receive tofacitinib tablet twice daily for 5 days under fasting conditions.
  Interventions: Drug: Tofacitinib
- Part 2: Treatment EF (JNJ-64251330) (Experimental): Participants will receive a single dose of JNJ-64251330 (dose 2), on Day 1 once under fasting conditions (Treatment E) in Period 1 followed by a single dose of JNJ-64251330 (dose 2), on Day 1 once with high fat breakfast (Treatment F) in Period 2. There will be a minimum of 5 days washout between dosing in the two treatment periods.
  Interventions: Drug: JNJ-64251330
- Part 2: Treatment FE (JNJ-64251330) (Experimental): Participants will receive a single dose of JNJ-64251330 (dose 2), on Day 1 once with high fat breakfast (Treatment F) in Period 1 followed by a single dose of JNJ-64251330 (dose 2), on Day 1 once under fasting conditions (Treatment E) in Period 2. There will be a minimum of 5 days washout between dosing in the two treatment periods.
  Interventions: Drug: JNJ-64251330

INTERVENTIONS:
Drug: JNJ-64251330 — JNJ-64251330 tablet will be administered orally.
  Arms: Part 1: Treatment A (JNJ-64251330); Part 1: Treatment B (JNJ-64251330); Part 1: Treatment C (JNJ-64251330); Part 2: Treatment EF (JNJ-64251330); Part 2: Treatment FE (JNJ-64251330)
Drug: Tofacitinib — Tofacitinib tablets will be administered orally.
  Arms: Part 1: Treatment D (JNJ-64251330)

SUMMARY:
The purpose of this study is to evaluate: systemic and local gut (rectum and sigmoid colon) exposure to JNJ-64251330, local tissue Pharmacodynamics (PD) using gut (rectum and sigmoid colon) biopsies (Part 1) and the effect of food on the rate and extent of absorption of JNJ-64251330 from oral tablet dosed with or without food (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI; weight [kilogram {kg}]/height^2 [meter {m}]^2) between 18.0 and 30.0 kilograms per meter square (kg/m^2) (inclusive), and body weight not less than 50.0 kg
* 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function, including: QTc interval less than or equal to (<=) 450 milliseconds (ms) for men and <= 470 ms for women
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, lipid panel, hematology, coagulation or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Have participant-reported normal consistency, regular bowel movements
* A woman must have a negative highly sensitive serum (beta-human chorionic gonadotropin [hCG])

Exclusion Criteria:

* History of hepatic or renal insufficiency; significant cardiac, vascular, pulmonary, endocrine, hematologic, rheumatologic, neurologic, oncologic, or psychiatric disease, or metabolic disturbances or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Active or chronic infection, a nontuberculous mycobacterial infection, or opportunistic infection (example, pneumocystosis and aspergillosis)
* History of severe allergic reaction to midazolam
* Contraindications to the use of tofacitinib per summary of product characteristics (SmPC)^14/ local prescribing information
* Female participant who is a breastfeeding mother

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Observed Plasma Concentrations (Cmax) of JNJ-64251330 | Predose, 0.25 hour (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h Postdose on Day 1 and Day 5; Predose on Day 2
  Cmax is maximum observed plasma concentrations during a dosing interval.
Part 1: Trough Observed Plasma Concentration (Ctrough) of JNJ-64251330 | Predose, 24 hour (h) Postdose on Day 5
  Ctrough is observed plasma concentration immediately prior to dosing on Day 5 and 24 h after last dose.
Part 1: Area Under the Plasma Concentration-Time Curve from 0 to 24 Hour (AUC [0-24 h]) of JNJ-64251330 | Predose, 0.25 hour (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 14 h, 24 h Postdose on Day 1 and Day 5; Predose on Day 2
  AUC (0-24 h) is defined as area under the plasma concentration-time curve from time 0 to 24 hours postdose will be evaluated.
Part 1: Area Under the Plasma Concentration-Time Curve from Time 0 to Time of Last Quantifiable Concentration (AUC [0-Last]) of JNJ-64251330 | Predose, 0.25 hour (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 14 h, 24 h Postdose on Day 1 and Day 5; Predose on Day 2
  AUC (0-Last) is defined as area under the plasma concentration versus time curve from time 0 to time of the last quantifiable concentration will be evaluated.
Part 1: Biopsy Gut (Rectum and Sigmoid Colon) Tissue Concentration of JNJ-64251330 | Day 6
  Biopsy gut (rectum and sigmoid colon) tissue concentration of JNJ-64251330 will be measured using liquid chromatography-mass spectrometry/mass spectrometry (LC MS/MS) assay method to evaluate systemic and local gut (rectum and sigmoid colon) exposure to JNJ-64251330.
Part 1: Change from Baseline in Levels of Phosphorylated Signal Transducer and Activator of Transcription (pSTATs) and other Pan-Janus kinase (JAK) Biomarkers | Baseline up to Day 6
  Change from baseline in levels of pSTATs and other JAK biomarkers in gut (rectum and sigmoid colon) biopsies as a function of compound and dose will be measured to evaluate local tissue pharmacodynamics (PD).
Part 2: Maximum Observed Plasma Concentrations (Cmax) of JNJ-64251330 | Predose, 0.25 hour (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h Postdose on Day 1; 24 h, 32 h, 36 h Postdose on Day 2; 48 h Postdose on Day 3
  Cmax is maximum observed plasma concentrations during a dosing interval.
Part 2: Time to achieve Maximum Observed Plasma Concentration (Tmax) of JNJ-64251330 | Predose, 0.25 hour (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h Postdose on Day 1; 24 h, 32 h, 36 h Postdose on Day 2; 48 h Postdose on Day 3
  Tmax is the maximum observed plasma concentration.
Part 2: Area Under the Plasma Concentration-Time Curve from Time 0 to 24 Hour (AUC [0-24 h]) of JNJ-64251330 | Predose, 0.25 hour (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h Postdose on Day 2
  AUC (0-24 h) defined as area under the plasma concentration-time curve from time 0 to 24 hour postdose will be evaluated.
Part 2: Area Under the Plasma Concentration-Time Curve from Time 0 to Time of Last Quantifiable Concentration (AUC [0-Last]) of JNJ-64251330 | Predose, 0.25 hour (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h Postdose on Day 1; 24 h, 32 h, 36 h Postdose on Day 2; 48 h Postdose on Day 3
  AUC (0-Last) defined as area under the plasma concentration versus time curve from time 0 to time of the last quantifiable concentration will be evaluated.
Part 2: Area Under the Plasma Concentration-Time Curve from Time 0 to Infinite Time (AUC [0-Infinite]) of JNJ-64251330 | Predose, 0.25 hour (h), 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h Postdose on Day 1; 24 h, 32 h, 36 h Postdose on Day 2; 48 h Postdose on Day 3
  AUC (0-Infinite) defined as area under the analyte concentration versus time curve from time 0 to infinite time will be evaluated.

SECONDARY OUTCOMES:
Parts 1 and 2: Incidence of Adverse Events (AEs) | Up to 35 days (Part 1); Up to 39 days (Part 2)
  Incidence of AEs will be evaluated to assess the safety and tolerability of JNJ 64251330 and tofacitinib. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product.
Parts 1 and 2: Number of Participants with Severity of AEs | Up to 35 days (Part 1); Up to 39 days (Part 2)
  Severity assessment for an AE will be completed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE Version 5.0). Severity grades ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening or Disabling and Grade 5= Death.
Part 1: Ratio of Gut (Rectum and Sigmoid colon) to Systemic Exposure | Up to Day 6
  Ratio of gut (rectum and sigmoid colon) to systemic exposure will be evaluated to assess the relative exposure of JNJ-64251330 versus tofacitinib.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Ma X, Borzillo G, Kothe MJC, Sanga M, Chu G, Greger JG, Deiteren A, Attiyeh E. A Phase I, Randomized, Multi-Dose Study to Evaluate the Enteric Selectivity and Safety of JAK Inhibitor, Lorpucitinib, in Healthy Participants. Clin Pharmacol Ther. 2024 May;115(5):1075-1084. doi: 10.1002/cpt.3170. Epub 2024 Jan 29. PMID 38159266